CLINICAL TRIAL: NCT03312803
Title: Mini-autogenous Skin Grafts With Skin Homografts Versus Autogenous Skin Graft for Covering Post Burn Wounds in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah El Din Mohamed Hassan, Resident doctor, Assiut University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Assiut
Record Dates: First submitted 2017-09-13; First posted 2017-10-18 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mini autogenous skin grafts (Active Comparator): we take the autogenous skin graft from the same patient then cut it into small pieces then we spread it over the burn wound on one limb then cover these small pieces with homogenous skin graft taken from another person.
  Interventions: Procedure: Mini autogenous skin graft
- Autogenous skin graft (Active Comparator): we take the regular autogenous one piece skin graft from the same patient and cover the burn wound on the other limb then we make a comparison between both limbs
  Interventions: Procedure: Mini autogenous skin graft

INTERVENTIONS:
Procedure: Mini autogenous skin graft — mini-autogenous skin grafts and skin homograft versus autogenous skin grafts for covering post burn wounds in children.

SUMMARY:
A prospective study comparing the use of mini-autogenous skin grafts and skin homograft versus autogenous skin grafts for covering post burn wounds in children.

DETAILED DESCRIPTION:
A prospective study comparing the use of mini-autogenous skin grafts and skin homograft versus autogenous skin grafts for covering post burn wounds in children so that the patient can continue on his/her normal life early with less deformities

ELIGIBILITY:
Inclusion Criteria:

* This study will include children (3-12) years old with (10-30) % body surface area burns, admitted to Assuit university hospital burn unit.
* The raw areas in both upper and lower limbs will be the site of the study.

Exclusion Criteria:

* Patients younger than 3 years old.
* Patients with burns more than 30% of total body surface area.
* Patients with medical or mental diseases.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
The major outcome is to specify if the regular single piece autogenous skin graft is better than the new technique that uses small pieces mini autogenous skin grafts for treatment of post burn wounds in children. or vice versa? | 2 years
  the spread of the small pieced autogenous skin grafts that are covered with homogenous skin graft over post burn wounds in children may give better results than the regular single pieced autogenous skin graft

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed St Salah El Din, Resident, Study Chair — Doctor Mostafa El Sonbaty
Locations (1):
- Assiut University Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Plan to do the study then share this study to be useful for all Plastic surgeons all around the world